CLINICAL TRIAL: NCT02775188
Title: interACTION: A Portable Joint Function Monitoring and Training System to Supplement Home Exercise Programs Following Anterior Cruciate Ligament Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of technical and feasibility issues with InterACTION, the study to investigate the system for individuals following ACL reconstruction was terminated.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, James J. Irrgang, PhD, PT, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO16020108
Record Dates: First submitted 2016-05-14; First posted 2016-05-17 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Therapy with InterACTION (Experimental): After ACL Reconstruction, subjects will undergo physical therapy 1 time per week supplemented by home exercise program with InterACTION device.
  Interventions: Device: interACTION
- Physical Therapy (Other): After ACL Reconstruction, subjects will undergo physical therapy 1 time per week
  Interventions: Other: Standard of Care Physical Therapy

INTERVENTIONS:
Device: interACTION
  Arms: Physical Therapy with InterACTION
Other: Standard of Care Physical Therapy
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to ascertain if home-based therapy with monitoring via telemedicine can overcome many barriers to compliance and improve rehabilitation following ACL reconstruction. Patients undergoing ACL Reconstruction will be followed for 6 weeks during their outpatient physical therapy treatment. Subjects will undergo weekly physical therapy or weekly physical therapy paired with InterACTION.

ELIGIBILITY:
Inclusion Criteria:

1. Between 15 to 30 years of age;
2. Have undergone ACL Reconstruction;
3. Being referred for post-operative outpatient physical therapy;
4. Agree to and able to perform pre-designed exercises that they would normally perform in a physical therapy program after ACL Reconstruction.

Exclusion Criteria:

1. Patients undergoing concomitant meniscal repair or other surgical procedure requiring modification of post-operative physical therapy program;
2. Patients with BMI >40 at the time of surgery;
3. Individuals who are not free of any other co-disability or comorbidity that would specifically impede disallow or otherwise hinder performance of physical therapy exercises;

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Value evaluated by the ratio of patient outcomes to costs of rehabilitation | 6 weeks
  Value will be evaluated by the ratio of patient outcomes to costs of rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States